CLINICAL TRIAL: NCT04120662
Title: Effectiveness of Shockwave Treatment for Proximal Fifth Metatarsal Stress Fracture in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Garcia Cugat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REHA-2019-02
Record Dates: First submitted 2019-07-25; First posted 2019-10-09 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Stress Fracture Metatarsal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Surgery group (Active Comparator): Surgical procedure according to the injury type
  Interventions: Procedure: Intramedullary screw fixation
- Goup B: Shockwave group (Active Comparator): 3 weekly sessions of Focused Shock Wave Treatment (F-ESWT), using an electrohydraulic device set to an energy flux density (EFD) of 0.21 mJ/mm2 and 2000 impulses
  Interventions: Device: Focused Shock Wave Treatment

INTERVENTIONS:
Procedure: Intramedullary screw fixation — A Kirschner wire was introduced in the proximal tuberosity under anteroposterior and lateral fluoroscopic control, following the bone axis and passing through the fracture line; a cannulated compressor screw in a diameter between 45 - 55 mm in the more satisfactory position to achieve the optimal fragments compression.
  Arms: Group A: Surgery group
Device: Focused Shock Wave Treatment — 3 weekly session, one per week, of focused shock waves, using an electrohydraulic device.
  Arms: Goup B: Shockwave group

SUMMARY:
Fifth metatarsal stress fracture is a failure of a healthy metatarsal bone subject to repetitive microdamages. It has a high prevalence in soccer players and is classified as a high-risk stress fracture. Based on Torg classification, the treatment options may be conservative or surgical. The recent increase of evidences about Shock Wave Treatment in different bone pathologies, including stress fractures, suggests the possibility to use this conservative intervention option also in patients candidate for surgery. This randomized clinical trial included 18 soccer players diagnosed of proximal fifth metatarsal stress fracture, randomly matched in Surgery group and Shock Wave group. Patients of Surgery group were treated with intramedullary screw fixation; patients of Shock Wave group received 3 weekly sessions of Focused Shock Wave Treatment (F-ESWT), using an electrohydraulic device set to an energy flux density (EFD) of 0.21 mJ/mm2 and 2000 impulses. Patients of both groups were followed monthly until their return to play (RTP) using radiography, Visual Analogue Scale (VAS), Tegner Activity Level Scale and AOFAS score.

ELIGIBILITY:
Inclusion Criteria:

* Male soccer players, aged over 18 years.
* Diagnosis of proximal fifth metatarsal stress fracture, according to clinical signs and symptoms and to radiologic findings
* Fracture occurred during soccer practice
* Informed consent signed

Exclusion Criteria:

* To be under 18 years old
* Traumatic fracture
* Fracture occurred out of soccer practice
* Patients with metatarsal shaft, neck or head fracture
* Patients with contraindication to receive surgical treatment
* Patients with contraindication to receive shock wave treatment
* Patients that refuse the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of X-Ray | Follow up until recovery (maximum of 6 months)
  X-Ray study
Period until return to play | Follow up until recovery (maximum of 6 months)
  When the patient can start the previous to injury activity

SECONDARY OUTCOMES:
Evaluation of Visual Analogue Scale | Follow up until recovery (maximum of 6 months)
  Subjective evaluation of the pain intensity from 0 (non-existent paint) to 10 (maximum pain feeling)
American Orthopedic Foot and Ankle Score | Follow up until recovery (maximum of 6 months)
  Measures the results of the treatment for complex foot and ankle injuries that combines a patient informed and a specialist informed report. Scores range from 0 to 100, with a healthy midfoot receiving 100 point.
Evaluation of Tegner activity scale | Follow up until recovery (maximum of 6 months)
  Tegner activity scale grades the daily life activities and recreational and professional sports practice. A score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports >6 score can only be achieved if the person participates in recreational or competitive sport.

CONTACTS AND LOCATIONS:
Overall Officials: Montse Garcia, Study Chair — Fundación Garcia Cugat
Locations (1):
- Fundacion Garcia Cugat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No